CLINICAL TRIAL: NCT04987840
Title: A Multi-Center Diagnostic Stewardship Program to Improve Respiratory Culture Utilization in Critically Ill Children
Acronym: BrighT STAR
Status: Enrolling by invitation | Type: Observational
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: IRB00263269; K24AI141580 (NIH); R01HS028634 (AHRQ)
Record Dates: First submitted 2021-07-28; First posted 2021-08-03 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Ventilator Associated Pneumonia; Tracheobronchitis
Keywords: Diagnostic Stewardship; Pediatric; Respiratory Culture Test
MeSH Terms: conditions — Pneumonia, Ventilator-Associated

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of this study is to evaluate implementation of diagnostic stewardship programs as a strategy to safely reduce antibiotic use, and to generate evidence and tools to support dissemination of diagnostic stewardship programs to a large and diverse group of hospitals.

DETAILED DESCRIPTION:
The Bright STAR Collaborative, or Testing STewardship to reduce Antibiotic Resistance Collaborative, is a prospective multicenter quality improvement (QI) program with the goal of implementing diagnostic stewardship interventions to reduce bacterial culture use as a strategy to reduce antibiotic overuse. Investigators will use data collected by participating sites to determine whether reliable implementation of clinical practice guidelines for evaluation of patients can decrease antibiotic use in pediatric intensive care units. Investigators will perform a quasi-experimental study to compare outcome data in pre- and post- periods.

Greater than or equal to 10 institutions will participate in this collaborative. Participating institutions will develop and implement an evidenced-based clinical decision-making tool as part of their quality improvement (QI) program in their pediatric intensive care unit (PICU).

Specific Aim 1: Evaluate whether locally devised quality improvement programs focused on diagnostic stewardship of respiratory cultures lead to a reduction in respiratory cultures and antibiotic use.

Specific Aim 2: To determine whether these quality improvement initiatives are associated with unintended consequence of patient harm such as mortality, length of stay, readmissions, ventilator associated infections, sepsis and septic shock.

Variables: total respiratory culture rates, culture results, ICU length of stay, mortality rates, hospital and ICU readmission, cause of death, ventilator-associated infection/ventilator-associated condition rate, sepsis, septic shock.

Analysis: The analytic approach equates to estimating and comparing the respiratory culture incidence during the "baseline/pre-implementation" and "post-implementation" periods, using a generalized linear mixed model (GLMM) assuming a Poisson distribution for the monthly number of respiratory cultures with the monthly number of ventilator days as an offset. Similar analyses will be performed for secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Institutions that plan to develop and implement a quality improvement program to reduce respiratory culture use in their Pediatric ICUs

Exclusion Criteria:

* Institutions that do not plan to develop and implement a quality improvement program to reduce respiratory culture use in their Pediatric ICUs

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: ICU patient populations from units that develop and implement a quality improvement program to reduce respiratory culture use
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Respiratory Culture Rate | up to 42 months
  Rate of endotracheal aspirate cultures; Change in respiratory cultures per 100 ventilator-days per month

SECONDARY OUTCOMES:
Broad spectrum antibiotic use for ICU days >2 days | up to 42 months
  Over all use of broad spectrum antibiotics; Total antibiotic days per 1,000 patient days per quarter
New initiations - Broad spectrum antibiotic use for ICU days >2 days | up to 42 months
  Antibiotic days per 1,000 patient-days per month (antibiotic days starting on day 3 of ICU admission)
Mortality | up to 42 months
  Death per hospital total ICU admissions comparing pre and post-intervention periods
Length of ICU stay | up to 42 months
  Days in ICU; median number of days comparing pre and post-intervention periods
ICU readmission | up to 42 months
  Readmission to the ICU within 7 days of discharge. The coordinating center will measure the change in rate of readmission per total ICU admissions comparing pre and post-intervention periods
Hospital readmission | up to 42 months
  Readmission to hospital within 7 days of discharge. The coordinating center will measure the change in rate of hospital readmission comparing pre and post-intervention periods
ventilator associated infections | up to 42 months
  Defined by the following: Rate of ventilator associated infections episodes per 100 ventilator-days per month
Sepsis | up to 42 months
  defined by the following: International Classification of Diseases (ICD)-10 codes ; Admissions with ICD-10 coded sepsis per total ICU admissions
Septic shock | up to 42 months
  Defined by the following: ICD-10 codes; Admissions with ICD-10 coded septic shock per total ICU admissions

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Milstone, MD, MHS, Principal Investigator — Johns Hopkins University
Locations (8):
- United States (8):
  - Johns Hopkins Children's Center, Baltimore, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - Children's Minnesota Hospital, Minneapolis, Minnesota
  - Children's Hospital and Medical Center Omaha, Omaha, Nebraska
  - Cleveland Clinic Children's Hospital, Cleveland, Ohio
  - Le Bonheur Children's Hospital, Memphis, Tennessee
  - Monroe Carell Jr. Children's Hospital, Nashville, Tennessee
  - Dell Children's Medical Center, Austin, Texas